CLINICAL TRIAL: NCT02738827
Title: Diode Laser Treatment of Pta Low Grade Bladder Tumors in the Outpatient Department.
Brief Title: Diode Laser Treatment of Bladder Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gregers Gautier Hermann (Other)
Responsible Party: Sponsor-Investigator, Gregers Gautier Hermann, consultant urologist, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URU05
Record Dates: First submitted 2015-12-21; First posted 2016-04-14 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser treatment (Other): Intervention is diode laser treatment of bladder cancer through a cystoscope without sedation of the patient.
  Interventions: Procedure: Laser treatment

INTERVENTIONS:
Procedure: Laser treatment — Intervention is diode laser treatment of bladder cancer through a cystoscope in the outpatient department

SUMMARY:
Laser treatment of pTa low grade bladder tumours in the outpatient department

Number of Subjects/Centres Planned: 20 patients will be included in this study. The study will be performed at Department of Urology, Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark.

Primary Objective: To show that small pTa bladder tumours safely can be removed with diode laser in an outpatient department Secondary Objective: To evaluate the patients experience with the laser treatment using QOL questionaires (symptom evaluation) and Visual Analog Scale Score (pain evaluation).

DETAILED DESCRIPTION:
Laser treatment of pTa low grade bladder tumours in the outpatient department

Number of Subjects/Centres Planned: 20 patients will be included in this study. The study will be performed at Department of Urology, Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark.

Primary Objective: To show that small pTa bladder tumours safely can be removed with diode laser in an outpatient department Secondary Objective: To evaluate the patients experience with the laser treatment using QOL questionaires (symptom evaluation) and Visual Analog Scale Score (pain evaluation).

Study Design: Open prospective study in patients with recurrent pTa low grade bladder tumours.

All patients will have their bladder tumour removed using a diode laser. The treatment will take place in the outpatient department (OPD) without any pain treatment. Biopsy from the tumour will be obtained before the procedure. If the biopsy shows low grade non-invasive bladder tumour, flexible cystoscopy will be repeated one month later in the OPD. At both procedures biopsy will be taken from the laser treated area.

If the per-operative biopsy shows high grade or invasive tumour, the patient will be referred for a re-resection at the operating theatre during admittance to the urology ward.

The pain is valuated by a Visual Analogue Scale Score and filled out immediately after each procedure.

Treatment induced symptoms will be evaluated using a QOL questionnaire which the patient fills out one week after the laser treatment and one week after the cystoscopies.

Population: Patients with histologically confirmed pTa urothelial bladder tumours Number of Subjects: Twenty patients Selection of Subjects: Patients scheduled for a trans urethral resection of bladder tumour (TUR-B) less than 1,5 cm at the operating theatre under general anaesthesia and without concomitant therapy with anticoagulants as Marevan, Marcoumar, and the new anticoagulants as Pradaxa etc. will after informed consent be included in the study.

Equipment:

Diode laser Storz, SPIES Biopsy forceps, Storz

Key Dates:

Overall duration of the study: 6 months included 1 months follow up Efficacy and Safety Variables Primary Endpoint: proportion of patients where the bladder tumours are completely removed by one laser treatment.

Secondary Endpoints:

* Portion of general urinary problems and QOL after laser treatment compared to cystoscopy and biopsy in the OPD
* Pain at the laser treatment and the cystoscopy assessed by Visual Analog Scale (VAS) Score.

Statistical Methods and Planned Analysis: Non-parametric and descriptive statistics will be performed

Parameters in the case report form (CRF):

Bladder cancer diagnosis (pTa low grade)

* Age
* Sex
* Mapping of lesions in normal, Clara Chrome, Spectra A and B filter cystoscopy
* Histology of all suspicious lesions
* SEPARATE CYSTOSCOPYFORM for laser TUR-B and the two follow up cystoscopies
* The duration of the laser treatment
* Expected clearance after the laser TUR-B
* The visibility during the laser TUR-B
* Visual Analog Scale Score result (to measure pain when laser treatment is performed and biopsies are taken in the OPD)

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of pTa low grade urothelial bladder tumor
* Tumor < 1.5 cm
* < 6 tumors

Exclusion Criteria:

* Patients with porphyria
* Known hypersensitivity to Hexvix® or porphyrins
* Use of any anticoagulants
* Macroscopic hematuria
* Pregnant or breast feeding women
* Expected poor compliance
* Patients < 18 years
* Patients who do not read or understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Tumour clearance | 1 month
  No bladder tumor tissue in biopsies obtained from areas where a bladder tumor one month earlier has been removed by use of diode laser.

CONTACTS AND LOCATIONS:
Overall Officials: Gregers G Hermann, MD, Principal Investigator — Dept Urology, Herlev/Gentofte hospital, Copenhagen, Denmark
Locations (1):
- Urological department, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No